CLINICAL TRIAL: NCT03623490
Title: Optimizing the Management of Patients With Oral Therapy: a Randomized Trial Evaluating the Impact of Management on the Occurrence of Side Effects
Brief Title: Optimizing the Management of Patients With Oral Therapy
Acronym: IPAC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Following an insufficient recruitment, the sponsor decided to halt prematurely inclusions
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IPAC
Record Dates: First submitted 2018-07-13; First posted 2018-08-09 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Kidney Cancer; Breast Cancer
Keywords: kidney cancer; breast cancer; oral therapy; managment
MeSH Terms: conditions — Kidney Neoplasms; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- accented follow-up (Experimental): Initial consultation with a trio oncologist / pharmacist / nurse; weekly telephone follow-up with a nurse between each treatment and follow-up visit with the oncologist at each renewal of treatment.
  Interventions: Other: managment of oral therapy
- standard follow-up (No Intervention): Initial consultation with the oncologist and follow-up visit with the oncologist

INTERVENTIONS:
Other: managment of oral therapy — Initial consultation with a trio oncologist / pharmacist / nurse
  Arms: accented follow-up

SUMMARY:
Oral anticancer treatments account a quarter of cancer treatments. These oral treatments are allowed at home, avoid hospitalization and limit the use of central venous routes. Oral treatments cause many side effects and patients are reluctant to report them because they are afraid that their treatment will be changed. But when these side effects are poorly managed, they can reduce adherence to treatment.

The main hypothesis of this randomized study is that the combination of an initial consultation with a trio (nurse, doctor, pharmacist) and a weekly telephone nurse follow-up during the administration of oral anticancer treatments decreases the rate and duration of side effects.

The main objective is to evaluate the impact at 3 months of a optimized management by an initial consultation with a trio nurse, doctor, pharmacist and a weekly nurse telephone follow-up versus a standard management on the level of digestive, skin and mucosal side effects of grade 3 in patients with oral chemotherapy.

This randomized study is realized in patients with kidney or breast cancer.

DETAILED DESCRIPTION:
Oral anticancer treatments account a quarter of cancer treatments. These oral treatments are allowed at home, avoid hospitalization and limit the use of central venous routes. Oral treatments cause many adverse effects (nausea, vomiting, digestive disorders, skin and mucous ...) that can significantly impact the quality of life. Patients are reluctant to report side effects because they are afraid that their treatment will be changed. But if these side effects are poorly managed, they can reduce adherence to treatment. The majority of devices are evaluated post-treatment and none relates to the treatment administration period.

The main hypothesis of this randomized study is that the combination of an initial consultation with a trio (nurse, doctor, pharmacist) and a weekly telephone nurse follow-up during the administration of treatments decreases the rate and duration of digestive, cutaneous and mucosal side effects.

The main objective is to evaluate the impact at 3 months of a optimized management by an initial consultation with a trio nurse, doctor, pharmacist and a weekly nurse telephone follow-up versus a standard management on the level of digestive, skin and mucosal side effects of grade 3 in patients with oral chemotherapy (Xeloda® or Sutent®).

ELIGIBILITY:
Inclusion Criteria:

1. Patient over 18 years old.
2. Men or women with kidney cancer treated with Sutent® chemotherapy (Cohort 1) according to the following schedule: 42-day course: 28 days of treatment + 14 days of break therapeutic)
3. Women with breast cancer treated with Xeloda® (Cohort 2) chemotherapy according to the following schedule: 21-day course: 14 days of treatment + 7 days of therapeutic break).
4. Patient (e) able to understand French read, write, speak.
5. Patient who received information about the study.
6. Written and signed consent.
7. Affiliation to a social security scheme.
8. Patient reachable by phone.

Exclusion Criteria:

1. Patient under guardianship, curatorship or safeguard of justice.
2. Patient with severe mental retardation impairing comprehension abilities.
3. Impossibility of submitting to the medical follow-up of the test.
4. If hospitalized at the time of inclusion: hospitalization forecast greater than 1 week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

PRIMARY OUTCOMES:
Rate of side effects | 6 months
  Side effects evaluated: digestive, cutaneous and mucosal grade 3 and 4

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Georges François Leclerc, Dijon, France